CLINICAL TRIAL: NCT00437060
Title: A Study of Neurocognitive Function in Children Treated for ALL
Brief Title: Brain Function in Young Patients Receiving Methotrexate for Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL06N1; NCI-2009-00315 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000528920; AALL06N1 (Other: Childrens Oncology Group); AALL06N1 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Childhood B Acute Lymphoblastic Leukemia; Childhood T Acute Lymphoblastic Leukemia; Cognitive Side Effects of Cancer Therapy; Long-Term Effects Secondary to Cancer Therapy in Children; Neurotoxicity Syndrome; Psychological Impact of Cancer; Untreated Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — Mental Status and Dementia Tests; Diffusion Tensor Imaging; Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and cerebrospinal fluid

GROUPS / COHORTS (1):
- Ancillary/Correlative (neurocognitive assessment, biomarkers)): Patients complete neurocognitive tests to assess thinking, memory, attention, and concentration. The baseline test is administered during the consolidation phase of chemotherapy and further tests are done at 1 year from baseline and 1 year after* the completion of study therapy.
  Patients undergo blood and cerebrospinal fluid collection periodically for biomarker, genotypic polymorphisms, and pharmacokinetic analysis. Patients undergo MRI diffusion-tensor imaging to correlate imaging with neuropsychological outcomes.
  Interventions: Procedure: Cognitive Assessment; Procedure: Diffusion Tensor Imaging; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Procedure: Psychosocial Assessment and Care

INTERVENTIONS:
Procedure: Cognitive Assessment — Ancillary studies
Procedure: Diffusion Tensor Imaging — Correlative studies
  Other Names: DTI
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Procedure: Psychosocial Assessment and Care — Ancillary studies
  Other Names: Psychosocial Assessment; Psychosocial Care; Psychosocial Care/Assessment; Psychosocial Studies; Psychosocial Support

SUMMARY:
This clinical trial is looking at brain function in young patients receiving methotrexate for acute lymphoblastic leukemia. Learning about the long-term effects of methotrexate on brain function may help doctors plan cancer treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the neuropsychological function in children with acute lymphoblastic leukemia treated with either high-dose methotrexate or escalating-dose methotrexate in the absence of cranial radiation and nelarabine.

II. Identify host polymorphisms that predict an increased risk of neurocognitive dysfunction or acute neurotoxicity in these patients.

III. Correlate neuropsychological outcome measures and the occurrence of acute neurotoxicity with host polymorphisms in these patients.

IV. Measure concentrations of 5-methyltetrahydrofolate, homocysteine, Ado, S-adenosylmethionine, S-adenosylhomocysteine, and other potentially relevant compounds in serum and cerebrospinal fluid during interim maintenance therapy with low- or high-dose methotrexate regimens, respectively, and correlate these endpoints with the occurrence of acute neurologic toxicity and long-term neurocognitive dysfunction in these patients.

V. Determine whether or not diffusion tensor imaging will identify areas of selective vulnerability in CNS and provide an imaging modality that predicts and/or correlates with neuropsychological outcome.

OUTLINE: This is a prospective, cohort, multicenter study.

Patients complete neurocognitive tests to assess thinking, memory, attention, and concentration. The baseline test is administered during the consolidation phase of chemotherapy and further tests are done at 1 year from baseline and 1 year after* the completion of study therapy.

Patients undergo blood and cerebrospinal fluid collection periodically for biomarker, genotypic polymorphisms, and pharmacokinetic analysis. Patients undergo MRI diffusion-tensor imaging to correlate imaging with neuropsychological outcomes.

NOTE: * Within 8 months to 24 months after the completion of study therapy for patients on AALL0232.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute lymphoblastic leukemia
* Enrolled on COG-AALL0434 (Cohort #1 only) or COG-AALL0232 (Cohorts #1 and #2)

  * Patients must have received either high-dose methotrexate or escalating-dose methotrexate during interim maintenance.
* No CNS-3 disease
* Patients must enroll within 8-24 months after completion of therapy on COG-AALL0232 and no evidence of relapsed or secondary malignancy
* No known significant neurodevelopmental disability unrelated to cancer diagnosis including, but not limited to, any of the following:

  * Down syndrome
  * Fragile X mental retardation
  * Autism
  * Pervasive developmental disability
  * Seizure disorder
* Attention-deficit hyperactivity disorder or specific learning disability (e.g., dyslexia) allowed
* No sensory impairment (e.g., pre-existing uncorrectable vision impairment or deafness)
* No cranial radiation therapy

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with newly diagnosed acute lymphoblastic leukemia meeting other criteria.
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2007-01; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in neurocognitive function by the Pediatric Quality of Life (PedQL) battery, Full Scale Intelligence Quotient (FSIQ) score | From baseline to up to 24 months
  Vocabulary and Block Design, subtests of the Wechsler Preschool and Primary Scale of Intelligence (WPPSI-III), Wechsler Children Intelligence Scale (WISC-IV) and Wechsler Adult Intelligence Scale (WAIS-III) (based on age) will be used to estimate FSIQ, using the tables provided by Sattler.
Polymorphisms as predictors of neurocognitive dysfunction or acute neurotoxicity | Up to 24 months

SECONDARY OUTCOMES:
Correlation between neuropsychological outcomes and acute neurotoxicity | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Winick, Principal Investigator — Children's Oncology Group
Locations (111):
- United States (101):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Southern California Permanente Medical Group, Downey, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Winthrop University Hospital, Mineola, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (3):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Hospital for Sick Children, Toronto, Ontario
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch